CLINICAL TRIAL: NCT05917158
Title: An Open-label, Single-arm Study to Evaluate the Efficacy and Safety of RC48-ADC Combined with JS001 in Postoperative Adjuvant Treatment of HER2-positive Upper Tract Urothelial Carcinoma (UTUC)
Brief Title: A Study of RC48-ADC Combined with JS001 for Postoperative Adjuvant Treatment of Upper Tract Urothelial Carcinoma
Acronym: 1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022DZKY-106-02
Record Dates: First submitted 2023-06-15; First posted 2023-06-23 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-07

CONDITIONS: Carcinoma; Upper Tract Urothelial Carcinoma; UTUC
MeSH Terms: conditions — Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RC48-ADC and JS001 (Experimental)
  Interventions: Drug: RC48-ADC and JS001

INTERVENTIONS:
Drug: RC48-ADC and JS001 — Patients in group will receive 6 x 3 week cycles of RC48-ADC (Disitamab Vedotin) 2mg/kg in combination with JS001 (Toripalimab) 3mg/kg intravenously, followed by toripalimab (3 mg/kg) every 3 weeks for up to 1 year.

SUMMARY:
This study will evaluate the efficacy and safety of intravenous RC48-ADC combined with JS001 in postoperative adjuvant therapy for HER2-positive upper tract urothelial carcinoma.

DETAILED DESCRIPTION:
This is an open-label, single-arm clinical trial to evaluate the efficacy and safety of RC48-ADC, a recombinant humanized anti-HER2 monoclonal antibody-Monomethyl auristatin E (MMAE) conjugate, in combination with JS001, a PD-1 monoclonal antibody, for the postoperative adjuvant treatment of HER2-positive upper tract urothelial carcinoma after radical nephroureterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* ≥18 years of age
* Post radical nephro-ureterectomy for upper tract tumour with predominant TCC component-squamoid differentiation or mixed TCC/SCC is permitted.
* Histologically confirmed TCC staged pT2-pT4 pN0-2 M0 or pTany N1-2 M0 (providing all grossly abnormal nodes are resected).
* Pathological tissue immunohistochemistry HER2 2~3+
* Fit and willing to receive adjuvant therapy with first cycle to be commenced within 90 days of radical nephro-ureterectomy if allocated
* ECOG(Eastern Cooperative Oncology Group) performance is 0~2.
* Available for long-term follow-up

Exclusion Criteria:

* Evidence of distant metastases
* Pure adenocarcinoma, squamous cell carcinoma or small cell or other variant histology
* Un-resected macroscopic nodal disease
* Concurrent muscle invasive bladder cancer (patients with concurrent Non-muscle invasive bladder cancer (NMIBC) will be eligible)
* Significant co-morbid conditions that would interfere with administration of protocol treatment
* Pregnancy; lactating women or women of childbearing potential unwilling or unable to use adequate non-hormonal contraception (male patients should also use contraception if sexually active);
* Previous malignancy in the last 5 years except for previous NMIBC, adequately controlled non melanoma skin tumours, CIS of cervix or LCIS of breast or localised prostate cancer in patients who have a life expectancy of over 5 years upon trial entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 5 years
  5-year Disease-free survival

SECONDARY OUTCOMES:
Overall survival (OS) | Patients followed-up for 5 years
  5-year Overall Survival
Metastasis free survival (MFS) | Patients are followed up for 5 years
  5-year Metastasis free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, China, Nanjing, Jiangsu, China